CLINICAL TRIAL: NCT01599429
Title: Use of FLT-TEP Scan as Predictive Marker and Early Prognostic in Patients Suffering From AML Treated by Chemotherapy
Brief Title: Study of the Predictive Marker FLT in Patients Suffering From AML
Acronym: TEP-FLT-LMA
Status: Withdrawn | Type: Observational
Why Stopped: No participants enrolled
Sponsor: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Responsible Party: Principal Investigator, Dr Éric E Turcotte, MD, Principal Investigator, Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Other Study IDs: CIMS-2011-01
Record Dates: First submitted 2011-11-04; First posted 2012-05-16 (Estimated); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML / LMA
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Positron emission tomography uses various radioactive tracers to measure the metabolic activity in a none-invasive way, and specially to follow the activity of the disease during the treatments.

Among those new tracers, fluorothymidine (18F-FLT) arouses a lot of interest. This new tool would allow to image and follow time wise acute myeloid leukemia (AML). The investigators want, with the (18F-FLT), to characterise the aggressivity of the tumors and the prognostic before and after chemotherapy treatment.

The aim of this study is to be able to identify earlier the responders, because if they are detected sooner, these patients will benefit from more aggressive treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years or above at the time of inclusion;
2. Patients newly diagnosed with acute myeloid leukemia;
3. No contraindication or intolerance to any of the components of the standard chemotherapy by induction (7+3);
4. Patients able to give written informed consent.

Exclusion Criteria:

1. Patients unable to tolerate decubitus position for at least 45 minutes;
2. Any previous neoplasia or other neoplasia simultaneously;
3. Previously treated buy radiotherapy, with bone marrow in the field of radiation;
4. Other chemotherapy treatment than the standard chemotherapy by induction (7+3), before the second FLT-TEP was done.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients newly diagnosed with acute myeloid, between October 2011 and October 2013, at the Centre Hospitalier Universitaire de Sherbrooke (CHUS).
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-10-31; Primary Completion 2017-10-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
To mesure the pronostic value of metabolic activity in the bone marrow with FLT-PET prior to chemotherapy in patients with AML disease. | September 2015

CONTACTS AND LOCATIONS:
Overall Officials: Éric E Turcotte, MD, Principal Investigator — Université de Sherbrooke, Centre Hospitalier Universitaire de Sherbrooke, Centre d'imagerie moléculaire de Sherbrooke (CIMS), Centre de recherche Étienne Le-Bel; Rami Kotb, MD, Principal Investigator — Université de Sherbrooke, Centre Hospitalier Universitaire de Sherbrooke
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada